CLINICAL TRIAL: NCT00359606
Title: Phase I Trial of 5-Fluoro-2'-Deoxycytidine With Tetrahydrouridine
Brief Title: 5-Fluoro-2'-Deoxcyctidine and Tetrahydrouridine to Treat Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 98127; PHI-16 (Other: California Cancer Consortium); UM1CA62505 (Other Grant/Funding Number: National Cancer Institute); NCI-2015-00655 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 06-C-0221 (Other: National Cancer Institute); NCT00378807 (obsolete NCT alias)
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Neoplasms
Keywords: DNA Methylation; Advanced Cancer; Methyltransferase Inhibitor; Epigenetics; Gene Re-Expression
MeSH Terms: conditions — Neoplasms | interventions — 5-fluoro-2'-deoxycytidine; Tetrahydrouridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (5-fluoro-2-deoxycytidine, tetrahydrouridine) (Experimental): Patients receive tetrahydrouridine PO on day 1; 5-fluoro-2-deoxycytidine PO on days 1 and 8; tetrahydrouridine IV over 3 hours on days 2-5, 8, and 9-12; and 5-fluoro-2-deoxycytidine IV over 3 hours on days 2-5 and 9-12 of course 1. For all subsequent courses, patients receive tetrahydrouridine IV over 3 hours and 5-fluoro-2-deoxycytidine IV over 3 hours on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: 5-Fluoro-2-Deoxycytidine (FdCyd); Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Tetrahydrouridine (THU)

INTERVENTIONS:
Drug: 5-Fluoro-2-Deoxycytidine (FdCyd) — Given PO and IV
  Other Names: 5-FLUORO-2'-DEOXYCYTIDINE; 5-fluoro-2-deoxycytidine; FdCyd; Ro 5-1090
Other: Laboratory Biomarker Analysis — Correlative Studies
Other: Pharmacological Study — Correlative Studies
Drug: Tetrahydrouridine (THU) — Given PO and IV
  Other Names: Tetrahydrouridine; THU

SUMMARY:
This phase I trial studies the side effects and best dose of 5-fluoro-2-deoxycytidine when given together with tetrahydrouridine in treating patients with solid tumors that have spread to other places in the body and usually cannot be cured or controlled with treatment (advanced). Drugs used in chemotherapy, such as 5-fluoro-2-deoxycytidine and tetrahydrouridine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of 5-fluoro-2'-deoxycytidine (5-fluoro-2-deoxycytidine) (FdCyd) administered by intravenous (IV) infusion over three hours with concomitant infusion of 350 mg/m2 of tetrahydrouridine (THU).

II. To describe the toxicities of FdCyd co-infused with THU.

III. To obtain preliminary evidence of anti-tumor activity in patients treated with this combination.

IV. To evaluate the pharmacokinetics of FdCyd and THU when co-infused.

V. To evaluate the oral bioavailability of FdCyd when co-administered with THU.

VI. When feasible, to measure the relative levels of the messenger ribonucleic acid (mRNA)'s for thymidylate synthase, deoxycytidine kinase, deoxycytidylate (dCMP) deaminase and other relevant enzymes; and the methylation status of p16 and other genes relevant to neoplasia.

OUTLINE: This is a dose-escalation study of 5-fluoro-2-deoxycytidine. Patients receive tetrahydrouridine orally (PO) on day 1; 5-fluoro-2-deoxycytidine PO on days 1 and 8; tetrahydrouridine IV over 3 hours on days 2-5, 8, and 9-12; and 5-fluoro-2-deoxycytidine IV over 3 hours on days 2-5 and 9-12 of course 1. For all subsequent courses, patients receive tetrahydrouridine IV over 3 hours and 5-fluoro-2-deoxycytidine IV over 3 hours on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Advanced, histologically-confirmed neoplastic disease refractory to standard therapy or for which no standard therapy exists
* Karnofsky performance status of at least 60% and estimated survival of at least two months
* Serum creatinine =< 2.0 mg/dl or creatinine clearance >= 50 ml/min
* Absolute neutrophil count (ANC) >= 1,500/ul
* Platelets >= 125,000/ul
* Bilirubin =< 1.5 mg/dl
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) =< 3 times the upper limits of normal
* Prior antineoplastic therapy must have been completed at least four weeks prior to the patient's entry on this study, or patients must have recovered from any expected side effects of the prior therapy; there is no limit on the number of cycles of prior chemotherapy
* Patients must be ineligible for or have refused participation in higher priority institutional protocols
* Written, voluntary, informed consent of the patient must be obtained in compliance with institutional, state and federal guidelines
* Pregnant patients are INELIGIBLE; all patients of child-bearing potential, both male and female, must be advised to practice adequate contraception; premenopausal women must have a negative pregnancy test prior to entry on this study
* Patients with any non-malignant intercurrent illness (e.g. cardiovascular, pulmonary, or central nervous system disease) which is either poorly controlled with currently available treatment, or which is of such severity that the investigators deem it inappropriate to treat the patient on this protocol are INELIGIBLE
* Patients currently being treated for a severe infection or who are recovering from major surgery are INELIGIBLE until recovery is deemed complete by the investigators
* The presence of measurable disease is NOT required for this phase I study; if bidimensionally measurable disease is present, baseline measurements of up to 3 indicator lesions should be made no earlier than four weeks prior to the first cycle of chemotherapy; pleural effusions, ascites and bone metastases are not considered measurable
* Complete blood count (CBC), differential count, platelet count, and blood chemistries should be done no earlier than 72 hours prior to each cycle of chemotherapy
* Pretreatment tests should be done no earlier than two weeks prior to the first cycle of chemotherapy
* Priority for accrual will be given to patients with breast cancer due to the in vitro data suggesting potential activity for this disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 1999-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of 5-fluoro-2-deoxycytidine (FdCyd) when given with tetrahydrouridine (THU) determined by dose-limiting toxicities | 28 days
  MTD is defined as the highest dose tested in which < 33% of patients experienced dose limiting toxicity. The toxicities observed at each dose level will be summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity (by National Cancer Institute Common Toxicity Criteria version 2.0 and nadir or maximum values for the laboratory measures), time of onset (i.e., cycle number), duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects by dose and by cycle.
Survival | Time from registration to time of death due to any cause, assessed up to 13 years
  Survival and time to failure will be summarized with Kaplan-Meier plots to describe the outcome of patients treated on this protocol.
Time to treatment failure | Time from registration to the first observation of disease progression, death due to any cause, or early discontinuation of treatment, assessed up to 13 years
  Survival and time to failure will be summarized with Kaplan-Meier plots to describe the outcome of patients treated on this protocol.

OTHER OUTCOMES:
Levels of mRNA's of interest | Up to 13 years
  The relative levels of mRNA's of interest and other biochemical assessments will be tabulated and described. These levels will be compared with clinical response in an exploratory manner. However, the heterogeneity of the patient population and the small number of patients treated at each dose make formal statistical analysis of the molecular studies unlikely.
Pharmacokinetic parameters of 5-fluoro-2-deoxycytidine in combination with tetrahydrouridine | Baseline, 15 & 30 minutes, 1, 2, 4, 6, 9 hours on days 1 & 8; baseline, 15 & 30 minutes, 1, 2, 2.5 hours after infusion start & 15 & 30 minutes, 1, 2, 4, 6 hours after infusion end on day 2; baseline on days 3, 9, & 15; 2.5 hours after infusion on day 12
  The pharmacokinetic data will be analyzed using compartmental and non-compartmental models for each patient. The estimated parameters will be tabulated by dose level with summary statistics (means and standard deviations, or medians and ranges). If appropriate, summary statistics will also be provided for the entire group of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Morgan, MD, Principal Investigator — City of Hope Medical Center
Locations (4):
- United States (4):
  - City of Hope National Medical Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California, Davis Cancer Center, Sacramento, California
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Carter SK. Editorial: Large-bowel cancer-The current status of treatment. J Natl Cancer Inst. 1976 Jan;56(1):3-10. doi: 10.1093/jnci/56.1.3. No abstract available. PMID 1255749
- [Background] Doroshow JH, Multhauf P, Leong L, Margolin K, Litchfield T, Akman S, Carr B, Bertrand M, Goldberg D, Blayney D, et al. Prospective randomized comparison of fluorouracil versus fluorouracil and high-dose continuous infusion leucovorin calcium for the treatment of advanced measurable colorectal cancer in patients previously unexposed to chemotherapy. J Clin Oncol. 1990 Mar;8(3):491-501. doi: 10.1200/JCO.1990.8.3.491. PMID 2407810
- [Background] Keyomarsi K, Moran RG. Folinic acid augmentation of the effects of fluoropyrimidines on murine and human leukemic cells. Cancer Res. 1986 Oct;46(10):5229-35. PMID 2944577
- [Derived] Holleran JL, Beumer JH, McCormick DL, Johnson WD, Newman EM, Doroshow JH, Kummar S, Covey JM, Davis M, Eiseman JL. Oral and intravenous pharmacokinetics of 5-fluoro-2'-deoxycytidine and THU in cynomolgus monkeys and humans. Cancer Chemother Pharmacol. 2015 Oct;76(4):803-11. doi: 10.1007/s00280-015-2857-x. Epub 2015 Sep 1. PMID 26321472
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-C-0221.html